CLINICAL TRIAL: NCT00352690
Title: A Phase II Study of Radiation Therapy, Paclitaxel Poliglumex, and Carboplatin in Stage III Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety of patients
Sponsor: Washington University School of Medicine (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-1195
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — paclitaxel poliglumex; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (first 12 eligible patients) (Other): Paclitaxel poliglumex 135 mg/m2 IV on day 1 of each 21 day cycle for a total of 2 cycles.
  Carboplatin AUC=5 IV over 30 minutes on day 1 of each 21 day cycle for a total of 2 cycles.
  Thoracic radiation therapy starting day 1 consisting of 66 Gy delivered in 2 Gy daily fractions.
  Paclitaxel poliglumex 175 mg/m2 IV beginning 3-5 weeks after completion of radiation therapy on day 1 every 21 days for a total of 2 cycles.
  Carboplatin AUC=6 IV beginning 3-5 weeks after completion of radiation therapy on day 1 every 21 days for a total of 2 cycles.
  Interventions: Drug: Paclitaxel poliglumex; Drug: Carboplatin; Radiation: External beam radiation therapy
- Cohort 2 (remaining patients) (Experimental): Paclitaxel poliglumex 175 mg/m2 IV on day 1 of each 21 day cycle for a total of 2 cycles.
  Carboplatin AUC=5 IV over 30 minutes on day 1 of each 21 day cycle for a total of 2 cycles.
  Thoracic radiation therapy starting day 1 consisting of 66 Gy delivered in 2 Gy daily fractions.
  Paclitaxel poliglumex 175 mg/m2 IV beginning 3-5 weeks after completion of radiation therapy on day 1 every 21 days for a total of 2 cycles.
  Carboplatin AUC=6 IV beginning 3-5 weeks after completion of radiation therapy on day 1 every 21 days for a total of 2 cycles.
  Interventions: Drug: Paclitaxel poliglumex; Drug: Carboplatin; Radiation: External beam radiation therapy

INTERVENTIONS:
Drug: Paclitaxel poliglumex
  Other Names: Xyotax
Drug: Carboplatin
  Other Names: Paraplatin
Radiation: External beam radiation therapy

SUMMARY:
This study is intended to evaluate the role of paclitaxel poliglumex and carboplatin in the treatment of unresectable Stage III non-small cell lung cancer along with radiation therapy in a multi-institutional trial. Consolidation chemotherapy with paclitaxel poliglumex and carboplatin will follow the completion of chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented NSCLC, including squamous cell carcinoma, adenocarcinoma (including bronchoalveolar cell), and large cell anaplastic carcinoma (including giant and clear cell carcinomas).
* Eligible Disease Stages: Inoperable IIIA and Selected IIIB
* Local radiation oncologist must approve patient eligibility prior to entry on study.
* Patients must have measurable disease.
* Prior Therapy:

  * ≥ 2 weeks since formal exploratory thoracotomy.
  * No prior chemotherapy or radiation therapy for NSCLC.
* ECOG performance status 0-1
* Required Initial Laboratory Values (must be submitted within 16 days prior to registration):

  * Granulocytes ≥ 1,500/µl
  * Platelets ≥ 100,000/µl
  * Calculated Creatinine Clearance ≥ 20 cc/min
  * Bilirubin < 1.5 mg/dl
  * AST (SGOT) < 2 x ULN
  * INR > 0.8 < 1.2* *Values apply exclusively to patients not being treated with warfarin. Values for patients being treating with warfarin should fall within the following therapeutic range: > 2.0 < 3.0.

Exclusion Criteria:

* Currently active second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse.
* Pregnant or nursing because of significant risk to the fetus/infant.
* Age <18 years.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* No HIV-positive patients receiving combination anti-retroviral therapy. Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy
* One-second forced expiratory volume (FEV1) <50% or hemoglobin-corrected carbon monoxide diffusion capacity (DLCO) <50% of predicted, as measured within 21 days of study entry
* Symptoms of esophageal dysfunction (dysphagia, odynophagia, or inability to swallow solid food) within 4 weeks prior to study randomization. Patients must not require prophylactic placement of percutaneous enterogastrostomy (PEG) tube or other non-oral nutritional supplement methods
* Weight loss of > 10% in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, M.D., Principal Investigator — Washington University School of Medicine
Locations (8):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Rush University Medical College, Chicago, Illinois
  - University of Kansas, Lawrence, Kansas
  - University of Minnesota, Twin Cities, Minneapolis, Minnesota
  - University of Missouri, Columbia, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - SUNY Upstate Medical University, Syracuse, New York

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment to the study was opened on 04/05/2006 and enrollment to the study closed 06/30/2008.
Period: Overall Study
Arm/Group | Cohort 1 (First 12 Eligible Patients) | Cohort 2 (Remaining Patients)
Started | 10 | 0
Completed | 8 | 0
Not Completed | 2 | 0
Not completed — Determined to be ineligible | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (First 12 Eligible Patients) | Cohort 2 (Remaining Patients) | Total
Number analyzed (Participants) | 8 | 0 | 8
Age, Continuous [Median (Full Range); unit: years] | 69 [53 to 77] |  | 69 [53 to 77]
Gender [Count of Participants; unit: Participants]
  Female | 5 |  |
  Male | 3 |  |
Region of Enrollment [Number; unit: participants]
  United States | 8 |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Rate
Description: * OS = time from patient registration to death of all causes
  * Estimated using Kaplan Meier
Time Frame: 6 months
Population: Participants with unknown expiration dates were censored at the date of last clinical contact.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (First 12 Eligible Patients) | Cohort 2 (Remaining Patients)
Number analyzed (Participants) | 8 | 0
percentage of participants | 73 |

2. Secondary Outcome: Failure-free Survival (FFS) Rate
Description: * The time between patient registration and a failure event (progression, relapse, or death of all cause, whichever is first)
  * Estimated using Kaplan Meier
Time Frame: 6 months
Population: Participants with unknown event dates were censored at the date of last clinical contact.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (First 12 Eligible Patients) | Cohort 2 (Remaining Patients)
Number analyzed (Participants) | 8 | 0
percentage of participants | 44 |

3. Secondary Outcome: Failure-free Survival (FFS)
Description: The time between patient registration and a failure event (progression, relapse, or death of all cause, whichever is first)
Time Frame: Completion of follow-up (follow-up ranged from 3 months to 6 years)
Population: Participants with unknown event dates were censored at the date of last clinical contact.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (First 12 Eligible Patients) | Cohort 2 (Remaining Patients)
Number analyzed (Participants) | 8 | 0
months | 6 [3.5 to 10.4] |

4. Secondary Outcome: Response Rates
Description: Overall best response using RECIST 1.0
Time Frame: 4 years
Measure: Number; unit: participants
Arm/Group | Cohort 1 (First 12 Eligible Patients) | Cohort 2 (Remaining Patients)
Number analyzed (Participants) | 8 | 0
participants
  Complete response | 1 |
  Partial response | 5 |
  Progressive disease | 1 |
  Unknown | 1 |

5. Secondary Outcome: Incidence and Severity of Radiation-induced Esophagitis
Time Frame: 30 days following completion of treatment (approximately 114 days)
Population: Using CTCAE Version 3.0
Measure: Number; unit: participants
Arm/Group | Cohort 1 (First 12 Eligible Patients) | Cohort 2 (Remaining Patients)
Number analyzed (Participants) | 8 | 0
participants
  Grade 1 | 1 |
  Grade 2 | 3 |
  Grade 3 | 0 |
  Grade 4 | 0 |
  Grade 5 | 0 |

6. Primary Outcome: Overall Survival (OS)
Description: OS = time from patient registration to death of all causes
Time Frame: Completion of follow-up (follow-up ranged from 3 months to 6 years)
Population: Participants with unknown expiration dates were censored at the date of last clinical contact.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (First 12 Eligible Patients) | Cohort 2 (Remaining Patients)
Number analyzed (Participants) | 8 | 0
months | 10.4 [3.5 to 18.5] |

7. Secondary Outcome: Incidence and Severity of Radiation-induced Pneumonitis
Time Frame: 30 days following completion of treatment (approximately 114 days)
Population: Using CTCAE Version 3.0.
Measure: Number; unit: participants
Arm/Group | Cohort 1 (First 12 Eligible Patients) | Cohort 2 (Remaining Patients)
Number analyzed (Participants) | 8 | 0
participants
  Grade 1 | 1 |
  Grade 2 | 2 |
  Grade 3 | 1 |
  Grade 4 | 0 |
  Grade 5 | 0 |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of treatment through 30 days after completion of treatment (approximately 114 days)
Arm/Group | Cohort 1 (First 12 Eligible Patients) | Cohort 2 (Remaining Patients)
Serious Adverse Events (participants affected / at risk) | 5/8 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (First 12 Eligible Patients) (N=8) | Cohort 2 (Remaining Patients) (N=0)
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Death NOS (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Febrile neutropenia (Infections and infestations) | 1 | 0
Hypotension (Cardiac disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Leukocytes (WBC) (Investigations) | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Myoglobin (Investigations) | 1 | 0
Neutrophils (Investigations) | 3 | 0
PTT (Investigations) | 1 | 0
Radiation pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Respiratory failure (death) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Troponin (Cardiac disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (First 12 Eligible Patients) (N=8) | Cohort 2 (Remaining Patients) (N=0)
AST (Investigations) | 2 | 0
Alkaline phosphatase (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blurred vison (Eye disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Confusion (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia/heartburn (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Edema (General disorders) | 1 | 0
Elevated troponin (Cardiac disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 4 | 0
Fatigue (General disorders) | 6 | 0
Febrile neutropenia (Infections and infestations) | 1 | 0
Fever - no infection (General disorders) | 1 | 0
Flashing lights/floaters (Eye disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 8 | 0
Hemorrhage - gastritis (Gastrointestinal disorders) | 1 | 0
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 0
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Infection with grade 0-2 neutrophils (Infections and infestations) | 3 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Leukocytes (WBC) (Investigations) | 5 | 0
Lymphopenia (Investigations) | 6 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Mood alteration - anxiety (Psychiatric disorders) | 1 | 0
Mood alteration - depression (Psychiatric disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 0
Neuropathy (Nervous system disorders) | 2 | 0
Neutrophils (Investigations) | 5 | 0
Pain: other (General disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Phantom pain (General disorders) | 1 | 0
Platelets (Investigations) | 8 | 0
Radiation pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Puritis (Skin and subcutaneous tissue disorders) | 2 | 0
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Weight loss (Investigations) | 1 | 0

LIMITATIONS AND CAVEATS:
(3) grade 5 serious adverse events occurred and led to the study closing early for the safety of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes